CLINICAL TRIAL: NCT02435901
Title: ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION (HSCT) IN PATIENTS WITH HIGH RISK HEMOGLOBINOPATHIES LIKE SICKLE CELL DISEASE AND β-THALESSEMIA-MAJOR USING REDUCED INTENSITY CONDITIONING REGIMEN
Brief Title: HSCT For Patients With High Risk Hemoglobinopathies Using Reduced Intensity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08057
Record Dates: First submitted 2015-04-24; First posted 2015-05-06 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Sickle Cell Disease; Beta Thalassemia-Major
Keywords: Reduced Intensity Conditioning Regimen
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia | interventions — Alemtuzumab; fludarabine; Melphalan; Cyclosporine; Mycophenolic Acid; Tacrolimus; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Reduced Intensity Regimen (Experimental): Administration of reduced doses of alemtuzumab (Campath-IH) IV 3mg test dose on Day -20 followed by daily dose of 10mg/dose on Day -19 to Day -17 for patients <10yrs or a daily dose of 15mg/dose on Day -19 to Day -17 for patients > 10yrs. Fludarabine 35mg/m2 daily for 4 days on Day -7 to Day -4. Melphalan 70mg/m2 daily for 2 days on Day -3 and Day -2. On Day -1 Cyclosporine OR Tacrolimus will be initiated along with Mycophenolate Mofetil as a graft vs host disease prophylaxis. On Day 0 the Human Leukocyte Antigen (HLA) matched or mismatched Hematopoietic Stem Cells from either the related or unrelated donor will be infused.
  Interventions: Drug: alemtuzumab (Campath IH); Drug: Fludarabine; Drug: Melphalan; Drug: Cyclosporine; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Biological: Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: alemtuzumab (Campath IH) — Alemtuzumab (Campath IH) is given daily over first 4 days, Day -20 to Day -17
  Other Names: Campath-IH
Drug: Fludarabine — Fludarabine 35/m2 is given daily over 4 days on Day -7 to Day -4.
Drug: Melphalan — Melphalan 70mg/m2 is given daily over 2 days on Day -3 to Day -2.
Drug: Cyclosporine — Immunosuppressant to prevent graft vs host disease is given on Day -1 prior to stem cell infusion
Drug: Mycophenolate mofetil — Immunosuppressant to prevent graft vs host disease is given on Day -1.
Drug: Tacrolimus — Immunosuppressant to prevent graft vs host disease is given Day -1 prior to stem cell infusion
Biological: Hematopoietic Stem Cell Transplantation — Human Leukocyte Antigen (HLA) matched or mismatched; related or unrelated hematopoietic stem cells to be transplanted on Day 0.

SUMMARY:
This study will evaluate the use of reduced intensity conditioning regimen in patients with high risk hemoglobinopathy Sickle Cell and B-Thalassemia Major in combination with standard immunosuppressive medications, followed by a routine stem cell transplant in order to assess whether or not it is as effective as myeloablative high dose chemotherapy and transplant.

DETAILED DESCRIPTION:
Standard myeloablative regimens are toxic to non-hematopoietic tissue and are associated with treatment related mortality and morbidity (TRM). Preparative regimens that are not myeloablative are associated with a greatly decreased incidence of TRM. In addition to providing a less toxic regimen, the reduced intensity chemotherapy preparative regimen also remains immunosuppressive enough to allow donor engraftment. Recent report of non-myeloablative regimens which resulted in engraftment of allogeneic stem cell in hematological malignancies raises the possibility that this conditioning regimen might be useful in achieving engraftment in non hematological disorder.

In an effort to achieve stable engraftment with any suitable donor stem cell source and to minimize toxicity the investigators have developed a new reduced intensity conditioning regimen for high risk hemoglobinopathies with the main aim of significantly suppressing the recipient's immune system and facilitate engraftment.

Non-myeloablative or reduced-intensity immunosuppressive preparative regimens have achieved a stable, mixed chimerism engraftment and successful allogeneic bone marrow transplants.

ELIGIBILITY:
Inclusion Criteria:

* Patient Inclusion Criteria for Sickle Cell Disease
* Patients at least one year of age to less than or equal to 21 years of age with (Sickle Cell Disease-SS or Sickle Cell-S-β-Thalassemia and with one or more of the following disease complications:
* Development of stroke on chronic transfusion protocol.
* Allosensitization on chronic transfusion therapy
* Impaired neuropsychological function and abnormal MRI scan
* Abnormal Transcranial Doppler studies
* Acute chest syndrome (2 to 3 episodes of acute chest syndrome in last 3 to 4 years).
* Ferritin level < 1500 mg/ml
* Recurrent painful priapism; 3-4 episodes/year requiring intervention.
* Recurrent vaso-occlusive crisis of at least 3 to 4 episodes/year.
* Osteonecrosis of multiple bones with documented destructive changes.
* Signed informed consent
* Patients physically and psychologically capable of undergoing transplantation and a period of strict isolation.
* Ferritin < 1500
* Liver Iron Concentration < 6mg/g

Patient Inclusion Criteria for β Thalassemia major Patients less than or equal to 21 years of age with B- Thalassemia major on routine monthly transfusion protocol or with one or more of the following complications;

1. Hepatomegaly.
2. Liver biopsy revealing evidence of portal fibrosis as A) Mild B) Moderate
3. Ferritin level≤ 1500ng/ml
4. Liver Iron Concentration (LIC) < 6mg/g

Exclusion Criteria:

* Exclusion Criteria for Both Sickle Cell and β Thalassemia Major Patient
* HIV positive result confirmed by Western Blot.
* Pregnancy (Pregnancy testing for females of child-bearing age will be performed and those with a positive serum β-Human Chorionic Gonadotropin will be excluded) and lactating females.
* Creatinine greater than two times the upper limit of normal for the laboratory,
* Pulmonary disease with FVC, FEV1 or DLCO parameters < 50% predicted (corrected for hemoglobin) or stage 3 or 4 sickle lung disease.
* Cardiac insufficiency or coronary artery disease requiring treatment
* Active infection requiring systemic antibiotic therapy with antibacterial, antifungal or antiviral agents
* Lansky performance score <70%- (Appendix B)
* Acute hepatitis/biopsy evidence of cirrhosis.
* Pulmonary Hypertension

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2008-12; Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center of New York, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Outcome data to include study findings.

REFERENCES:
- [Derived] King AA, Kamani N, Bunin N, Sahdev I, Brochstein J, Hayashi RJ, Grimley M, Abraham A, Dioguardi J, Chan KW, Douglas D, Adams R, Andreansky M, Anderson E, Gilman A, Chaudhury S, Yu L, Dalal J, Hale G, Cuvelier G, Jain A, Krajewski J, Gillio A, Kasow KA, Delgado D, Hanson E, Murray L, Shenoy S. Successful matched sibling donor marrow transplantation following reduced intensity conditioning in children with hemoglobinopathies. Am J Hematol. 2015 Dec;90(12):1093-8. doi: 10.1002/ajh.24183. Epub 2015 Oct 6. PMID 26348869

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no significant events in the study which prevented participant enrollment.
Groups:
- Reduced Intensity Regimen: Administration of reduced doses of alemtuzumab (Campath-IH) IV 3mg test dose on Day -20 followed by daily dose of 10mg/dose on Day -19 to Day -17 for patients <10yrs or a daily dose of 15mg/dose on Day -19 to Day -17 for patients > 10yrs. Fludarabine 35mg/m2 daily for 4 days on Day -7 to Day -4. Melphalan 70mg/m2 daily for 2 days on Day -3 and Day -2. On Day -1 Cyclosporine OR Tacrolimus will be initiated along with Mycophenolate Mofetil as a graft vs host disease prophylaxis. On Day 0 the Human Leukocyte Antigen (HLA) matched or mismatched Hematopoietic Stem Cells from either the related or unrelated donor will be infused
  alemtuzumab (Campath IH): Alemtuzumab (Campath IH) is given daily over first 4 days, Day -20 to Day -17
  Fludarabine: Fludarabine 35/m2 is given daily over 4 days on Day -7 to Day -4.
  Melphalan: Melphalan 70mg/m2 is given daily over 2 days on Day -3 to Day -2.
  Cyclosporine: Immunosuppressant to prevent graft vs host disease is given on Day -1 prior to s
Period: Overall Study
Arm/Group | Reduced Intensity Regimen
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Reduced Intensity Regimen: Administration of reduced doses of alemtuzumab (Campath-IH) IV 3mg test dose on Day -20 followed by daily dose of 10mg/dose on Day -19 to Day -17 for patients <10yrs or a daily dose of 15mg/dose on Day -19 to Day -17 for patients > 10yrs. Fludarabine 35mg/m2 daily for 4 days on Day -7 to Day -4. Melphalan 70mg/m2 daily for 2 days on Day -3 and Day -2. On Day -1 Cyclosporine OR Tacrolimus will be initiated along with Mycophenolate Mofetil as a graft vs host disease prophylaxis. On Day 0 the Human Leukocyte Antigen (HLA) matched or mismatched Hematopoietic Stem Cells from either the related or unrelated donor will be infused.
  alemtuzumab (Campath IH): Alemtuzumab (Campath IH) is given daily over first 4 days, Day -20 to Day -17
  Fludarabine: Fludarabine 35/m2 is given daily over 4 days on Day -7 to Day -4.
  Melphalan: Melphalan 70mg/m2 is given daily over 2 days on Day -3 to Day -2.
  Cyclosporine: Immunosuppressant to prevent graft vs host disease is given on Day -1
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hemoglobinopathies [Count of Participants; unit: Participants] | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Cell Engraftment of Donor Cells
Description: Sustained stem cell engraftment of donor cells will be evaluated by chimerism (FISH fluorescence in situ hybridization OR VNTR (Variable Number of Tandem Repeats), based on recipient/donor gender, at 30 days, 100 days, 6 months and 1 year following the use of reduced intensity conditioning.
Time Frame: 1 year
Population: All 29 participants were analyzed at time-points of 30 days, 100 days, 6 month and 1 year for sustained stem cell engraftment of donor cells.
Measure: Count of Participants; unit: Participants
Groups:
- Reduced Intensity Regimen: Alemtuzumab (Campath-IH) IV 3mg test dose on Day -20 followed by 10mg/dose on Day -19 to Day -17 for patients <10yrs or a daily dose of 15mg/dose on Day -19 to Day -17 for patients > 10yrs. Fludarabine 35mg/m2 daily for 4 days on Day -7 to Day -4. Melphalan 70mg/m2 daily for 2 days on Day -3 and Day -2. Day -1 Cyclosporine OR Tacrolimus along with Mycophenolate Mofetil as a graft vs host disease prophylaxis. On Day 0 the HLA matched or mismatched Hematopoietic Stem Cells from either the related or unrelated donor will be infused.
  alemtuzumab (Campath IH): Alemtuzumab (Campath IH) is given daily over first 4 days, Day -20 to Day -17
  Fludarabine: Fludarabine 35/m2 is given daily over 4 days on Day -7 to Day -4.
  Melphalan: Melphalan 70mg/m2 is given daily over 2 days on Day -3 to Day -2.
  Cyclosporine: Immunosuppressant to prevent graft vs host disease is given on Day -1 prior to s
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 29
Participants | 29

2. Secondary Outcome: Assessment of Treatment Related Mortality and Morbidity
Description: Patients will be evaluated for incidence and severity of graft versus host disease, infection, and cardiopulmonary complications.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Reduced Intensity Regimen: Alemtuzumab (Campath-IH) IV 3mg test dose on Day -20 followed by daily dose of 10mg/dose on Day -19 to Day -17 for patients <10yrs or a daily dose of 15mg/dose on Day -19 to Day -17 for patients > 10yrs. Fludarabine 35mg/m2 daily for 4 days on Day -7 to Day -4. Melphalan 70mg/m2 daily for 2 days on Day -3 and Day -2. Day -1 Cyclosporine OR Tacrolimus along with Mycophenolate Mofetil as a graft vs host disease prophylaxis. On Day 0 the HLA matched or mismatched Hematopoietic Stem Cells from either the related or unrelated donor will be infused.
  alemtuzumab (Campath IH): Alemtuzumab (Campath IH) is given daily over first 4 days, Day -20 to Day -17
  Fludarabine: Fludarabine 35/m2 is given daily over 4 days on Day -7 to Day -4.
  Melphalan: Melphalan 70mg/m2 is given daily over 2 days on Day -3 to Day -2.
  Cyclosporine: Immunosuppressant to prevent graft vs host disease is given on Day -1 prior to s
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 29
Participants
  Grade I-Grade III GVHD | 13
  Chronic GVHD | 9
  No complications | 7

3. Secondary Outcome: Event Free Survival; Number of Participants Who Survived at 2 Years
Description: 29 participants will be evaluated for Event Free Survival.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 29
Participants
  Expired Secondary to Sepsis | 1
  Expired Secondary to GVHD | 2
  Survived Participants | 26

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to the end of the first year post transplant.
Description: Serious adverse events included 3 participants who expired within the first year post transplant. One participant expired secondary to sepsis episode. Two participants expired secondary to complications of Grade III-IV graft vs. host disease.
  Adverse event included13 patients experienced adverse event of Grade I-II graft vs host disease, and responded to oral and/or topical treatment.
Groups:
- Reduced Intensity Regimen: Alemtuzumab (Campath-IH) IV 3mg test dose on Day -20 followed by daily dose of 10mg/dose on Day -19 to Day -17 for patients <10yrs or a daily dose of 15mg/dose on Day -19 to Day -17 for patients > 10yrs. Fludarabine 35mg/m2 daily for 4 days on Day -7 to Day -4. Melphalan 70mg/m2 daily for 2 days on Day -3 and Day -2. Day -1 Cyclosporine OR Tacrolimus along with Mycophenolate Mofetil as a graft vs host disease prophylaxis. Day 0 the HLA matched or mismatched Hematopoietic Stem Cells from either the related or unrelated donor will be infused.
  alemtuzumab (Campath IH): Alemtuzumab (Campath IH) is given daily over first 4 days, Day -20 to Day -17
  Fludarabine: Fludarabine 35/m2 is given daily over 4 days on Day -7 to Day -4.
  Melphalan: Melphalan 70mg/m2 is given daily over 2 days on Day -3 to Day -2.
  Cyclosporine: Immunosuppressant to prevent graft vs host disease is given on Day -1
  Mycophenolate mofetil: Immunosuppressant to prevent graft vs host
Arm/Group | Reduced Intensity Regimen
All-Cause Mortality (participants affected / at risk) | 3/29
Serious Adverse Events (participants affected / at risk) | 3/29
Other Adverse Events (participants affected / at risk) | 13/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Intensity Regimen (N=29)
Graft vs Host Disease (Gastrointestinal disorders) | 2 (2) — 22 participants experienced various grades of graft vs host disease (GVHD), inclusive of skin & gut (acute and chronic). Of the 22, 2 participants expired from complication of graft vs host disease and 1 participant expired from a septic episode.
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced Intensity Regimen (N=29)
Grade I-II Graft vs Host Disease (Immune system disorders) | 13 — 13 patients experienced adverse event of Grade I-II graft vs host disease, and responded to oral and/or topical treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT02435901/Prot_SAP_000.pdf